CLINICAL TRIAL: NCT02381678
Title: A Retrospective Study to Collect the Data From the Patients Who Had the Perimount Heart Valve Replacement Surgery in China During 2001 to 2007
Status: Completed | Type: Observational
Sponsor: Edwards (Shanghai) Lifesciences Medical Supplies Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: Edwards-CN-001
Record Dates: First submitted 2015-03-05; First posted 2015-03-06 (Estimated); Results first posted 2016-10-17 (Estimated); Last update posted 2016-10-17 (Estimated); Status verified 2016-05

CONDITIONS: Mitral Valve or Aortic Valve Replacement
Keywords: Heart Valve Replacement; Perimount 2900; China; Perimount 6900P

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Subjects implanted with Perimount Heart Valve: Only one group was set for this study, including all enrolled subjects who implanted with Perimount Heart Valve during 2001 to 2007
  Interventions: Device: Perimount 2900/6900 Heart Valve

INTERVENTIONS:
Device: Perimount 2900/6900 Heart Valve — This is a retrospective study which ask the subjects implanted with Perimount Heart Valve during 2001 to 2007 back hospital for follow up visit.

SUMMARY:
The objective of the study is to obtain the clinical data from patients who had the Perimount Heat Valve (Type:6900P and 2900) Replacement Surgery in Guangdong General Hospital during 2001-2007 in order to evaluate the performace of this heart valve prothesis and collect the patients' post-operation infomation including the current living status, mortality rate, and the possibility of re-operation，bleeding and thrombosis.

This is a retrospective , observentional clinical study to be conducted in Guangdong General Hospital in China. This study will enroll up to 200 patients.

ELIGIBILITY:
Inclusion Criteria:

* The patients who implanted with Perimount Heart Valve (Type: 6900P and 2900) during 2001-2007 in Guangdong General Hospital in China
* The patients agree to join the study and sign the ICF

Exclusion Criteria:

* No specific exclusion criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The patients who had the Perimount Heart Valve (Type: 6900P and 2900) Replacement Surgery during 2001-2007 in Guangdong General Hospital in China
Sampling Method: Non-Probability Sample
Enrollment: 225 (Actual)
Dates: Start 2014-05; Primary Completion 2015-11 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Huiming Guo, M.D, Principal Investigator — Guangdong Provincial People's Hospital
Locations (1):
- Guangdong General Hospital, Guangzhou, Guangdong, China

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Investigators find total 253 patients who implanted Perimount Heart Valve during 2001 to 2007 in the Guangdong General Hospital. After the contact with these patients or their relatives, 225 patients agree to join the study.
Groups:
- Age Group Under 60 Years Old: 54 subjects implanted Perimount Heart Valve when the age was under 60.
- Age Group Between 60 and 70 Years Old: 139 subjects implanted Perimount Heart Valve when the age was between 60 and 70 years old (>=60,<70)
- Age Group Above 70 Years Old: 32 subjects implanted Perimount Heart Valve when the age was above 70
Period: Overall Study
Arm/Group | Age Group Under 60 Years Old | Age Group Between 60 and 70 Years Old | Age Group Above 70 Years Old
Started | 54 | 139 | 32
Completed | 54 | 139 | 32
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: This is one-arm study, all 225 subjects included in the Full Analysis Set.
Groups:
- All Patients Enrolled in Study: The whole group included 225 enrolled subjects. All 225 subjects included in the FAS(Full Analysis Set).
Arm/Group | All Patients Enrolled in Study
Number analyzed (Participants) | 225
Age, Continuous [Mean (Full Range); unit: years] | 63 [16 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 119
  Male | 106
Etiology of subjects [Number; unit: participants]
  Rheumatic | 124
  Degenerated | 51
  Endocardititis | 6
  Ischemic | 18
  Miscellaneous | 26
Preoperative Classification of NYHA assessment [Number; unit: participants] — The criteria for NYHA assessment listed below:
  Class I: Cardiac disease, but no symptoms and no limitation in ordinary physical activity, e.g. no shortness of breath when walking, climbing stairs etc.
  Class II: Mild symptoms (mild shortness of breath and/or angina) and slight limitation during ordinary activity.
  Class III: Marked limitation in activity due to symptoms, even during less-than-ordinary activity, e.g. walking short distances (20-100 m).
  Comfortable only at rest. Class IV: Severe limitations. Experiences symptoms even while at rest. Mostly bed-bound patients.
  participants
    Class I | 5
    Class II | 79
    Class III | 96
    Class IV | 31
    Not Known | 14
The numbers of valves implanted simultaneously [Number; unit: participants]
  Single Valve Replacement | 174
  Double Valves Replacement | 48
  Triple Valves Replacement | 3
The concomitant surgery [Number; unit: participants]
  Coronary Artery Bypass Grafting | 41
  Left Atrial Reduction | 5
  Tricuspid valvuloplasty | 75
  Radiofrequency Ablation | 4
The time for Extracorporeal Circulation and Cross Clamp in surgery [Mean (Standard Deviation); unit: minutes]
  Time for Extracorporeal Circulation | 137.9 (66.6)
  Time for cross clamp | 89.5 (40.2)

OUTCOME MEASURES:

1. Primary Outcome: The Performance Evaluation of Perimount Heart Valve(Type:6900P and 2900) by Echocardiography
Description: This is a one-arm study. All enrolled 225 subjects are required to be back Gungdong General Hospital to do an Echocardiography
Time Frame: 7-15 years after heart valve replacement surgery (during 2001-2007)
Measure: Number; unit: Percentage of all subjects
Groups:
- One-arm Group Included All Enrolled Subjects: This group included total 225 enrolled participants
Arm/Group | One-arm Group Included All Enrolled Subjects
Number analyzed (Participants) | 225
Percentage of all subjects
  Freedom from SVD at 5 years | 100
  Freedom from SVD at 10 years | 54.54
  Freedom from SVD at 15 years | 26.51
  Overall survival rate at 5 years | 81.33
  Overall survival rate at 10 years | 62.41
  Overall survival rate at 15 years | 51.63

ADVERSE EVENTS:
Time Frame: All patients implanted with Perimount Heart Valves during 2001 to 2007. And investigators collect these patients' current healthy information and report the safety and efficacy results of a 9-15 year follow-up investigation
Description: The serious adverse events for these subjects included death and reoperation. And the adverse events mainly included SVD (structure of valve deterioration)
Arm/Group | Age Group Under 60 Years Old | Age Group Between 60 and 70 Years Old | Age Group Above 70 Years Old
Serious Adverse Events (participants affected / at risk) | 12/54 | 60/139 | 22/32
Other Adverse Events (participants affected / at risk) | 14/54 | 27/139 | 2/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Age Group Under 60 Years Old (N=54) | Age Group Between 60 and 70 Years Old (N=139) | Age Group Above 70 Years Old (N=32)
Death (Cardiac disorders) | 8 (8) | 56 (56) | 22 (22)
Re-operation (Cardiac disorders) | 4 (4) | 4 (4) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Age Group Under 60 Years Old (N=54) | Age Group Between 60 and 70 Years Old (N=139) | Age Group Above 70 Years Old (N=32)
SVD (Cardiac disorders) | 14 (14) | 27 (27) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No